CLINICAL TRIAL: NCT03724786
Title: Management of Pregnancies With Suspected Preeclampsia Based on 6-hour Versus 24-hour Urine Protein Collection - a Randomized Double Blind Controlled Pilot Study
Brief Title: Management of Suspected Preeclampsia Based on 6-hour Versus 24-hour Urine Protein Collection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Hadas Ganer Herman, Principal Investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0168-18-WOMC
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calculated collection (Experimental): Patients in this arm will collect urine for protein for 6 hours, and then an additional 18 hours. The result of the 6-hour collection will be multiplied by four, and the result will serve as the "calculated collection", for pregnancy management. The additional 18 hour collection will serve for: 1. Patient blinding. 2. Calculation of the total 24-hour protein collection for reference.
  Interventions: Diagnostic Test: Six-hour urine protein collection
- Control collection (No Intervention): Patients in this arm will collect urine for protein for 6 hours, and then an additional 18 hours. The result of the total 24-hour collection will serve for pregnancy management. The initial 6-hour collection will serve for patient blinding.

INTERVENTIONS:
Diagnostic Test: Six-hour urine protein collection — This intervention includes the analysis of a 6-hour urine collection for protein, to serve for a calculated 24-hour result, according to which pregnancy will be managed.
  Arms: Calculated collection

SUMMARY:
In this trial - the investigators plan to study the efficacy of pregnancy management in cases of suspcted preeclampsia, based on a 6-hour urine collection for protein, as compared to the standard 24-hour collection. For participants hospitalized at the maternal fetal unit at our institution, one sample of urine collected over 6 hours will be analyzed, and a second one following an additional 18 hours. Participants will be blinded to the urine collection result used to manage their pregnancy (actual 24 hour collection versus calculated 24-hour collection), as will be their attending physicians. An external physician will compare the two urine collection results, and in case only one is pathological (>300 mg), will notify the research team and the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the Edith Wolfson Medical Center for suspected preeclampsia, for whom hospitalization was recommended for urine collection for protein and blood pressure follow up
* Gestational age >24+0 weeks and < 42+0 weeks
* Consent to participation

Exclusion Criteria:

* Patients with features of severe preeclampsia at presentation - blood pressure >160/110, headache, blurred vision, right upper quadrant pain, liver transaminase abnormality, increased creatinine level, thrombocytopenia.
* Patients whom were decided to be delivered (regardless of protein collection)
* Multiple gestation
* Chronic hypertension
* Pre-gestational diabetes mellitus
* Thrombophilia (APLA)
* Intrauterine growth retardation
* Lack of prenatal care

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with an adverse maternal outcome composite | Up to 18 weeks
  Defined as one of the following maternal complications - hepatic or renal injury, placental abruption, eclampsia, thrombocytopenia, cerebral morbidity, respiratory morbidity, blood pressure > 160/110, need for anti-hypertensives

SECONDARY OUTCOMES:
Number of participants whose neonate had an adverse neonatal outcome composite | Up to 18 weeks
  Defined as one of the following neonatal complications - respiratory distress syndrome, necrotizing enterocolitis, mechanichal ventilation, phototherapy, neonatal intensive care unit admission, sepsis, death
Gestational age | Single evaluation, up to 18 weeks from recruitment
  Gestational age at delivery
Number of patients who underwent a cesarean delivery | Single evaluation, up to 18 weeks from recruitment
  Delivery by cesarean surgery
Number of patients who underwent labor induction | Single evaluation, up to 18 weeks from recruitment
  Need for labor induction, by mechanichal or pharmaceutical means

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Ganer Herman, MD, Principal Investigator — Obstetrics and Gynecology, Edith Wolfson Medical Center
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herman HG, Barda G, Miremberg H, Gonen N, Torem M, Kleiner I, Bar J, Weiner E. Management of pregnancies with suspected preeclampsia based on 6-hour vs 24-hour urine protein collection-a randomized double-blind controlled pilot trial. Am J Obstet Gynecol MFM. 2021 Sep;3(5):100429. doi: 10.1016/j.ajogmf.2021.100429. Epub 2021 Jun 25. PMID 34182189